CLINICAL TRIAL: NCT01178463
Title: Spermatogonial Stem Cells in Azoospermic Patients: a Comparison Between Obstructive and Non-obstructive Azoospermia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Adrian Ellenbogen, Hillel Yaffe Medical Center
Other Study IDs: HYMC-0065-09
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- I. Obstructive Azoospermia
  Interventions: Other: Biospecimen staining
- II. Non-Obstructive Azoospermia Patients
  Interventions: Other: Biospecimen staining

INTERVENTIONS:
Other: Biospecimen staining — The sections will be incubated with rabbit anti GPR125 followed by Cy3-conjugated anti rabbit secondary antibodies.
  Groups: I. Obstructive Azoospermia
Other: Biospecimen staining — The sections will be incubated with rabbit anti GPR125 followed by Cy3-conjugated anti rabbit secondary antibodies.
  Groups: II. Non-Obstructive Azoospermia Patients

SUMMARY:
The researchers hypothesized that nonobstructive azoospermia might be associated with a reduction OF SSCs in seminiferous tubules as compared with obstructive azoospermia. Testicular sperm specimens that had been previously extracted from azoospermic patients will be paraffin embedded and stained with anti GPR-125. After antigen retrieval, the sections will be incubated with rabbit anti GPR125 followed by Cy3-conjugated anti rabbit secondary antibodies. Those found to be SSCs will be counted using light microscopy, and compared between patients with obstructive (n=11) and non-obstructive azoospermia (n=9).

ELIGIBILITY:
Inclusion Criteria:

* Azoospermic patients

Exclusion Criteria:

* Patients with sperm cells

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infertile male patients treated at the Hillel Yaffe Medical Center IVF Unit
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
SSCs were identified in both obstructive and nonobstructive azoospermia patients. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center - IVF Unit, Hadera, Israel